CLINICAL TRIAL: NCT04399369
Title: Preventing Early Childhood Caries with Silver Diamine Fluoride - a 12-month Randomised Clinical Trial
Brief Title: Preventing Caries with Silver Diamine Fluoride
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chun Hung Chu, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20200520
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: 5% NaF and 38% SDF
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SDF (Experimental): 38% silver diamine fluoride solution
  Interventions: Device: SDF
- NaF (Active Comparator): 5% sodium fluoride varnish
  Interventions: Device: NaF

INTERVENTIONS:
Device: SDF — 38% silver diamine fluoride solution
  Arms: SDF
Device: NaF — 5% sodium fluoride varnish
  Arms: NaF

SUMMARY:
Background: Early childhood caries (tooth decay, ECC) affected 55% 5-year-old Hong Kong children, and 70% of these children had gross destruction of the upper anterior teeth with negative long-term impacts on health and quality of life. The existing standard of care for prevention of ECC, topical application of 5% sodium fluoride (NaF) varnish, is inadequate. In Hong Kong and other parts of the world, 38% silver diamine fluoride (SDF) solution, applied topically to cavities, is used to arrest ECC. Work published by our research group suggests it likely also has a preventive effect of ECC. Moreover, SDF has been shown to be preventive in tooth decay in permanent teeth. Nevertheless, no pivotal clinical trial has been performed to support a change in usual practice.

Aim: This is a Phase II single-centre randomized, double-blind, active-controlled, parallel-group pragmatic trial with two arms to assess the effectiveness of 38% SDF and 5% NaF in preventing new caries lesions in primary anterior teeth. Methods: 688 three-year-old kindergarten children who are healthy will be recruited, stratified by school, and block randomized to receive either 38% SDF (treatment group) or 5% NaF (standard treatment group) therapy on primary upper anterior teeth. This sample size is sufficient for a superiority trial with power at 90%, allowing for a 15% dropout rate. The primary outcome is the number of sound tooth surfaces that become cavitated caries per child at 12-month follow-up. The secondary outcome is the number of carious tooth surfaces developed after baseline that become arrested at 12-month for each child. Dental examinations for the status of caries (active or arrested) will be conducted by the same calibrated examiner. The examiner, children and children's parents will be blind to treatment allocation. Parents will be surveyed to study the children's oral health-related behaviours and socioeconomic backgrounds, which will allow the adjustment for effect modification. Possible results and implications: If the results are as anticipated, it will help change the standard of care for caries prevention. If adopted in Hong Kong, SDF therapy will prevent 20,800 (13% of the 160,000) kindergarten children from having caries developed in their anterior teeth, thus reduce significantly the burden of ECC of the children and related stress of their family. Moreover, the results will be widely available and increase adoption of SDF in other countries to reduce the global burden of ECC among children.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy, with parental consents

Exclusion Criteria:

* uncooperative and difficult to manage, have major systemic diseases such as porphyria, or are on long-term medication such as anti-epileptic drugs.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 688 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
caries prevention | at 12-month follow-up
  the number of sound tooth surfaces that become cavitated caries per child

CONTACTS AND LOCATIONS:
Locations (1):
- Local kindergartens, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng FM, Yan IG, Duangthip D, Lo ECM, Gao SS, Chu CH. Caries Prevention Using Silver Diamine Fluoride: A 12-Month Clinical Trial. Int Dent J. 2023 Oct;73(5):667-673. doi: 10.1016/j.identj.2022.12.005. Epub 2023 Jan 20. PMID 36682908
- [Derived] Gao SS, Zheng FM, Chen KJ, Duangthip D, Lo ECM, Chu CH. Comparing two fluoride therapies for caries management in young children: study protocol for a randomised clinical trial. Trials. 2021 Aug 4;22(1):519. doi: 10.1186/s13063-021-05496-y. PMID 34348775